CLINICAL TRIAL: NCT02892006
Title: LOL: It's All Improv After Cancer! The Impact of Improvisational Comedy on Well-Being Among Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Arash Asher, MD, Director, Cancer Survivorship & Rehabilitation, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00045372
Record Dates: First submitted 2016-08-11; First posted 2016-09-08 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Distress; Breast Neoplasms; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants in the study will participate a 6 week improv intervention.
  Interventions: Behavioral: Improvisational Comedy

INTERVENTIONS:
Behavioral: Improvisational Comedy — 6 week curriculum in improvisational comedy. Each class meets for 1.5 hours for 6 consecutive weeks.

SUMMARY:
Managing distress and improving well-being is critically important for optimal survivorship care. Treatment of distress leads to better adherence to treatment, better communication, fewer calls and visits to the oncologist's office, and avoidance of development of severe anxiety or depression. Based on national guidelines, distress is typically managed with pharmacologic options (i.e. benzodiazepines), support groups, individual counseling, or chaplaincy services. To our knowledge, the role of a structured improvisational comedy (improv) program in reducing distress and improving well-being has never been evaluated in the oncology setting.

DETAILED DESCRIPTION:
With over 14 million cancer survivors today in the United States comes a unique constellation of challenges and opportunities for health care providers trying to optimize health at a time when many patients are struggling and open to learning new skills for strengthening their own resiliency and ability to cope. Not only does a significant subset of patients with cancer experience an increase in negative emotions, such as distress, anxiety and depression, but they often also experience a lack of positive emotions (Hart 2010). Managing distress and improving well-being is critically important for optimal survivorship care. Treatment of distress leads to better adherence to treatment, better communication, fewer calls and visits to the oncologist's office, and avoidance of development of severe anxiety or depression (Partridge, Wang et al. 2003; Carlson and Bultz 2004; 2014). Based on national guidelines, distress is typically managed with pharmacologic options (i.e. benzodiazepines), support groups, individual counseling, or chaplaincy services. To our knowledge, the role of a structured improvisational comedy (improv) program in reducing distress and improving well-being has never been evaluated in the oncology setting.

ELIGIBILITY:
Inclusion Criteria:

* Female, diagnosed with breast cancer stage 1-3 (no distant metastases)
* Completed cancer treatment (including chemotherapy, radiation therapy, biologic treatment, and/or any combination) at least 1 month (30 days) from their last treatment and no more than 12 months (365 days) post-treatment. Long term hormonal/biologic treatments are ok.
* Female age ≥ 18
* Scores a at least 4/10 (≥4) on the National Comprehensive Cancer Network Distress Thermometer
* Agrees to complete study surveys
* Agrees to attend 6 improv classes
* English speaking
* Emotionally stable (per physician clearance) to participate in this series

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Feasibility | Baseline to 6 weeks after baseline
  We will define feasibility by our attrition rate. We will assess the rate of accrual and the number of patients who complete the intervention

SECONDARY OUTCOMES:
Symptoms | Baseline to 6 weeks after baseline (t1); one month after t1
  We will assess the impact of a 6-week improv program on patient reported symptoms using the PROMIS-29 scale.
Well Being | Baseline to 6 weeks after baseline (t1); one month after t1
  We will assess the impact of a 6-week improv program on well being. Well-being will be assessed using the FACT-G scale.
Loneliness | Baseline to 6 weeks after baseline (t1); one month after t1
  We will assess the impact of a 6-week improv program on loneliness. Loneliness will be assessed using the UCLA Loneliness Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Asher, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No